CLINICAL TRIAL: NCT06295185
Title: How Social Ventures Boost Performance and Sustain Businesses With Digital Therapeutic Workplace Technology (Smartphone App 'Maro') Designed to Support Individual Employee's Mental Health
Brief Title: Digital Therapeutic Workplace Technology as a Employee Management Tool and Employee's Mental Health Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Chang Hyung Hong, Principal Investigator, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AJOUIRB-IV-2024-097
Record Dates: First submitted 2024-02-16; First posted 2024-03-06 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Depression; Mental Health Issue
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mental health treated with digital intervention app 'Maro' (Experimental): Intervention group will use 'Maro app' which was developed to improve mental health for 8weeks.
  Through 8weeks intervention group will record their status more than once a day and utilize specific functions in the app.
  They will also have meetings once a week in the online chat in order to share their own experience about Maro application use with other employees in the same branch.
  Interventions: Other: application MARO
- Digital Sham App (Sham Comparator): Control group will use Sham app for 8weeks.
  Interventions: Other: Sham application

INTERVENTIONS:
Other: application MARO — It is a mental healthcare application aim to improve mental health.
  Arms: mental health treated with digital intervention app 'Maro'
Other: Sham application — It is a sham application in order to control spill over bias.
  Arms: Digital Sham App

SUMMARY:
The purpose of the study is to determine whether a digital healthcare app for employee's mental health can effectively improve the mental health of Hisbeans's employees and the managerial performance of Hisbeans, which is represented as a 'social enterprise'.

DETAILED DESCRIPTION:
Hisbeans is a social enterprise where employees are consist of individual with mental disabilities.

'Hisbeans' employees(N = 150 subjects) will be randomly assigned to Group 1 (maro intervention), or Group 2 (control app intervention) by cluster randomization depending on the branch of the company.

* MARO intervention group: MARO (mental health digital application) use
* Control group: sham app use

The intervention period will be 8weeks.

ELIGIBILITY:
Inclusion Criteria:

1. HISBEANS store employees
2. Age: 18 years old or older
3. possessing a smartphone with internet connection
4. subjects agree to participate in the study

Exclusion Criteria:

1. Those who have symptoms of psychotic disorder are acutely active or advanced, making clinical intervention difficult
2. Those who has been started or changed their antidepressant medication within the last 1 month or cannot be maintained stably during the intervention period
3. Those who are non-literate
4. Those who have used the Maro app previously
5. Those who couldn't use Maro app in their own smartphone
6. Those who participate in another intervention study
7. Those who have a serious medical condition that prevents them from participating in the intervention and efficacy evaluation
8. Those who is unable to participate fully and cooperatively by the judgment of the researcher

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2024-05-20 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Change in network on the Standard Name Generator Approach scale | 4weeks, 8weeks after starting treatment
  * Description: A validated self-reported list of names assessing the subject's network scores
  * minimum and maximum values: from no name to the maximum available subject employees in the focal company that subject employees work for
  * score meaning: an individual subject generating more names means he or she has more connected people in the company
Change in depression symptoms severity on the Patient Health Questionnaire-9 | 4weeks, 8weeks after starting treatment
  * Description: Validated self-reported questionnaire assessing the severity of depression symptom
  * minimum and maximum values: 9-item scale with total scores between 0 and 27
  * score meaning: higher scores indicate greater symptoms severity

SECONDARY OUTCOMES:
Change in social capital on the Social Capital Scale | 4weeks, 8weeks after starting treatment
  * Description: Based on the validated self-reported name assessing the person's network scores, researchers calculate the inverse degree to which individuals hold less constraints in the network landscape
  * minimum and maximum values: a scale between 0 and 1 multiplied by the number of subjects individuals
  * score meaning: higher scores indicate greater social capital
Change in perceived workload on the Perceived Workload Scale | 4weeks, 8weeks after starting treatment
  * Description: Validated self-reported questionnaire assessing the complexity of jobs and the work-related stress
  * minimum and maximum values: a 4-item scale with total scores between 0 and 28
  * score meaning: higher scores indicate greater perceived workload
Change in job self-efficacy on the Job Self-Efficacy Scale | 4weeks, 8weeks after starting treatment
  * Description: Validated self-reported questionnaire assessing the efficacy of one's job and tasks
  * minimum and maximum values: a 11-item scale with total scores between 0 and 77
  * score meaning: higher scores indicate greater job self-efficacy
Change in sense of meaningfulness for job on the Sense of Meaningfulness for Job Scale | 4weeks, 8weeks after starting treatment
  * Description: Validated self-reported questionnaire assessing the sense of meaningfulness toward one's job
  * minimum and maximum values: a 6-item scale with total scores between 0 and 42
  * score meaning: higher scores indicate greater sense of meaningfulness for job
Change in work orientation toward his or her job on the Work Orientation Scale | 4weeks, 8weeks after starting treatment
  * Description: Validated self-reported questionnaire assessing one's work orientation toward his or her job
  * minimum and maximum values: categorical values among 'economic-value group', 'achievement group', and 'calling group'
  * score meaning: one sorting into a certain categorical value means one such
Change in sense of psychological safety on the Perception of Psychological Safety Scale of Company Employees | 4weeks, 8weeks after starting treatment
  * Description: Validated self-reported questionnaire assessing one's perception of psychological safety within the company
  * minimum and maximum values: a 7-item scale with average scores between 0 and 7
  * score meaning: higher scores indicate greater sense of psychological safety
Change in firm performance on the Company weekly sales records | 4weeks, 8weeks after starting treatment
  * Description: Validated objective measure of firm's performance assessing the department's weekly revenue
  * minimum and maximum values: a monetary scale between 0 and possibly generatable revenue during firm's operation time
  * score meaning: higher sales indicate greater firm performance
Change in amsenteeism/leaves on the absenteeism/leave scales for employees with severe mental disabilities | 4weeks, 8weeks after starting treatment
  * Description: Validated numeric, objective measure assessing the individual employees' absenteeism or turnover cases, among which we also measure the employees with severe mental disabilities.
  * minimum and maximum values: the number of individuals scale between 0 and the maximum possible employees working for the firm.
  * score meaning: higher number indicates greater amsenteeism/leaves
Change in stress regulation skill on the Emotional/Cognitive/Behavioral State Questionnaire | 4weeks, 8weeks after starting treatment
  * Description: self-reported questionnaire assessing stress regulation skill
  * minimum and maximum values: 3-item scale with total scores between 3 and 30
  * score meaning: higher scores indicate greater stress regulation skill
Change in anxiety symptoms severity on the General Anxiety Disorder-7items scale | 4weeks, 8weeks after starting treatment
  * Description: Validated self-reported questionnaire assessing the severity of anxiety symptom
  * minimum and maximum values: 7-item scale with total scores between 0 and 21
  * score meaning: higher scores indicate greater symptoms severity
Change in perceived stress level on the Perceived Stress Scale | 4weeks, 8weeks after starting treatment
  * Description: Validated self-reported questionnaire assessing perceived stress
  * minimum and maximum values: 10 scale with total scores between 0 and 40
  * score meaning: higher scores indicate greater perceived stress
Change in social functioning on Social Adaptation Self Rating Scale | 4weeks, 8weeks after starting treatment
  * Description: Validated self-reported questionnaire assessing social motivation and behavior
  * minimum and maximum values: 21-item scale with total scores between 21 and 84
  * score meaning: higher scores indicate greater social functioning
Change in positive psychological capital on Korean version of Positive Psychological Capital Scale | 4weeks, 8weeks after starting treatment
  * Description: Validated self-reported questionnaire assessing positive psychological capital, which consist of self-efficacy, hope, optimism, and resilience
  * minimum and maximum values: 18-item scale with total scores between 18 and 90
  * score meaning: higher scores indicate greater Positive Psychological Capital
Change in Organizational Companionship on Organizational Culture Inventory | 4weeks, 8weeks after starting treatment
  * Description: Validated self-reported questionnaire assessing Organizational Companionship
  * minimum and maximum values: 28-item scale with total scores between 28 and 196
  * score meaning: higher scores indicate a higher degress of organizational companionship
Change in individual's social network on Lubben Social Network Scale-18 | 4weeks, 8weeks after starting treatment
  * Description: Validated self-reported questionnaire assessing an individual's social network of relatives, friends, and neighbors.
  * minimum and maximum values: 18-item scale with total scores between 0 and 90
  * score meaning: higher scores indicate a larger social network

CONTACTS AND LOCATIONS:
Overall Officials: Chang Hyung Hong, Ph.D, Principal Investigator — Ajou Medical Center
Locations (1):
- Ajou Medical University, Suwon, South Korea

IPD SHARING:
Plan to Share IPD: No